CLINICAL TRIAL: NCT03857373
Title: Renal Cancer Detection Using Convolutional Neural Networks
Acronym: RCCCNN
Status: Recruiting | Type: Observational
Sponsor: Nessn Azawi (Other)
Responsible Party: Sponsor-Investigator, Nessn Azawi, Associate professor, Zealand University Hospital
Organization: Zealand University Hospital (Other)
Other Study IDs: Zealand_UCRU
Record Dates: First submitted 2019-02-26; First posted 2019-02-28 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Kidney Cancer
Keywords: Renal Cancer; Machine Learning
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Renal Cancer: Patients identified with RCC

SUMMARY:
We aim to experiment and implement various deep learning architectures in order to achieve human-level accuracy in Computer-aided diagnosis (CAD) systems. In particular, we are interested in detecting renal tumors from CT urography scans in this project. We would like to classify renal tumor to cancer, non cancer, renal cyst I, renal cyst II, renal cyst III and renal cyst VI, with high sensitivity and low false positive rate using various types of convolutional neural networks (CNN). This task can be considered as the first step in building CAD systems for renal cancer diagnosis. Moreover, by automating this task, we can significantly reduce the time for the radiologists to create large-scale labeled datasets of CT-urography scans.

DETAILED DESCRIPTION:
We aim to experiment and implement various deep learning architectures in order to achieve human-level accuracy in Computer-aided diagnosis (CAD) systems. In particular, we are interested in detecting renal tumors from CT urography scans in this project. We would like to classify renal tumor to cancer, non cancer, renal cyst I, renal cyst II, renal cyst III and renal cyst VI, with high sensitivity and low false positive rate using various types of convolutional neural networks (CNN). This task can be considered as the first step in building CAD systems for renal cancer diagnosis. Moreover, by automating this task, we can significantly reduce the time for the radiologists to create large-scale labeled datasets of CT-urography scans.

ELIGIBILITY:
Inclusion Criteria:

* All patient with RCC, who underwent surgery

Exclusion Criteria:

* Patients with RCC, who did not underwent surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with RCC
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Predicting recurrences | 5 years
  Predicting recurrences of RCC

CONTACTS AND LOCATIONS:
Locations (1):
- Zealand University Hospital, Roskilde, Denmark

IPD SHARING:
Plan to Share IPD: No